CLINICAL TRIAL: NCT06808776
Title: Stories to Prevent (StoP) HPV Cancers: A Communication Intervention to Increase HPV Vaccination Among Diverse Populations.
Brief Title: Stories to Prevent (StoP) HPV Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, William Calo, Associate Professor of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00025798
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Human Papillomavirus Vaccination; Emotions
Keywords: Human papillomavirus vaccine; Narrative communication; Emotions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer survivor narrative video (Experimental): Parents randomly assigned to this arm will receive the video intervention using their personal devices around two weeks before their child's wellness visit. The video will be approximately 4 minutes in length with three parts: (1) Cancer experience, (2) Vaccine recommendation, and (3) Closing message.
  Interventions: Other: Cancer survivor narrative
- Placebo video (Placebo Comparator): Parents randomly assigned to this arm will receive the placebo video using their personal devices around two weeks before their child's wellness visit. The placebo video is about healthy eating tips for families with children. The video will be approximately 4 minutes in length.
  Interventions: Other: Healthy eating tips

INTERVENTIONS:
Other: Cancer survivor narrative — The narrative video intervention has three parts: (1) Cancer experience - the cancer survivor narrates his/her experience with an HPV-related cancer, including diagnosis, treatment, and how cancer affected their personal life or family; (2) Vaccine recommendation - the cancer survivor provides brief information about the safety and effectiveness of the HPV vaccine and recommend that parents get the HPV vaccine for their child to prevent cancers; and (3) Closing message - The sentence "HPV vaccine is cancer prevention. Talk to your child's healthcare provider about getting the HPV vaccine during the next clinic visit" will appear on the screen.
  Arms: Cancer survivor narrative video
Other: Healthy eating tips — A publicly available video about healthy eating tips for families with children.
  Arms: Placebo video

SUMMARY:
This randomized controlled trial (RCT) evaluates the association of a narrative communication intervention on human papillomavirus (HPV) vaccination rates among 9- to 12-year-olds. The intervention is a brief video from local cancer survivors narrating their stories with an HPV-related cancer diagnosis and recommending the HPV vaccine for cancer prevention. RCT participants will be the parents (n=200) of children ages 9-12 who have not initiated HPV vaccination. Participants will be randomized (1:1) to our intervention or control (placebo video) one week before their child's next primary care visit. Our primary outcome is HPV vaccine initiation (first dose of the HPV vaccine series) among children ages 9-12 at the time of the wellness visit. The study also explores the effect of narratives on theory-based mediators of HPV vaccination, including parents' cognitive (e.g., risk perception) and emotional reactions (e.g., hope, anticipated regret).

DETAILED DESCRIPTION:
Despite the availability of the human papillomavirus (HPV) vaccine that can prevent over 37,300 HPV-related cancers in the US every year, only 62.6% of girls and boys were up-to-date in 2022. Low-quality provider recommendations and time constraints during clinic visits limit parents' opportunities to discuss and make HPV vaccination decisions. Pre-visit education to parents could complement provider communication to promote HPV vaccination. There is a critical need to identify better communication strategies to increase HPV vaccine uptake, including the use of narrative messaging and existing digital technologies in clinics and at home (electronic health records, patient portal, mobile devices). The Stories to Prevent (StoP) HPV Cancers Study is a randomized controlled trial (RCT) to evaluate the association of a narrative communication intervention delivered through digital and mobile technology before clinic visits on HPV vaccine initiation rates. A sample of 200 parents of unvaccinated children ages 9-12 will be randomized to receive our intervention or control (placebo video). Participants will be recruited from general pediatric and family medicine clinics affiliated with Penn State Health. We will also examine the effect of narrative communication on theory-based psychological mediators of HPV vaccine initiation and narrative communication processes, specifically parents' cognitive and emotional reactions.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian of a 9-12 year old receiving primary care at a Penn State Health clinic
* Their child has not previously received or initiated the HPV vaccine
* Is able to read and understand spoken English or Spanish
* Has a valid email address and access to a mobile phone, table, desktop or laptop computer to engage in the intervention

Exclusion Criteria:

* Parent of guardian is less than 18 years of age
* Unable to read and understand spoken English or Spanish
* Does not have access to a mobile phone, table, desktop or laptop computer

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine initiation, 9-12 year olds | One week after clinic visit
  The proportion of children ages 9-12 who have initiated HPV vaccination (first dose) during their scheduled clinic visit.

SECONDARY OUTCOMES:
HPV vaccine initiation stratified by age | One week after clinic visit
  The proportion of children ages 9-12 who have initiated HPV vaccination (first dose) by during their scheduled clinic visit stratified by age group (9-10 vs 11-12)
HPV vaccine initiation stratified by sex | One week after clinic visit
  The proportion of children ages 9-12 who have initiated HPV vaccination (first dose) during their scheduled clinic visit stratified by sex (male vs female)
HPV vaccine initiation stratified by race/ethnicity | One week after clinic visit
  The proportion of children ages 9-12 who have initiated HPV vaccination (first dose) during their scheduled clinic visit stratified by race/ethnicity (White, Black, Hispanic, Others)
HPV vaccine communication in clinics | One week after clinic visit
  Measure quality indicators of HPV vaccine recommendation, including the use of a presumptive announcement (i.e., noting the child's age, saying the child should get the vaccine today, using language that assumes the parent will accept the vaccine, focusing on disease prevention) and opportunities for the parent to voice concerns or questions and receive answers from the provider.
Believability | One week after the intervention
  Measure adapted from 12 items focusing on coverage, plausibility, completeness, and consistency with a 5-point scale (5=strongly agree to 1=strongly disagree)
Character identification | One week after the intervention
  Measure adapted from 6 items that use a 5-point scale focusing on similarity (5=strongly agree to 1=strongly disagree)
Health beliefs | One week after the intervention
  Measure adapted from 31 items focusing on risk susceptibility, severity, barriers, benefits, and self-efficacy rated on a 5-point scale (5=strongly agree to 1=strongly disagree)
Positive affect | One week after the intervention
  Measure adapted from 3 items on hope using a 5-point scale (5=strongly agree to 1=strongly disagree)
Negative affect | One week after the intervention
  Measure adapted from 9 items on negative affect using a 5-point scale (5=strongly agree to 1=strongly disagree)
Acceptability of digital health interventions | One week after the intervention
  Measure adapted from 10 items to assess acceptability of digital health interventions using 5-point scale (5=strongly agree to 1=strongly disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided